CLINICAL TRIAL: NCT01360970
Title: Hepatitis A Vaccination in Patients With Rheumatoid Arthritis Treated With TNF-inhibitors and/or Methotrexate
Brief Title: Hepatitis A Vaccine in Patients With Immunomodulating Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Rombo (Other)
Responsible Party: Sponsor-Investigator, Lars Rombo, Professor, Sormland County Council, Sweden
Organization: Sormland County Council, Sweden (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EU 2009-016055-22
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Response to Hepatitis A Vaccine
Keywords: hepatitis A vaccine; TNF-alfa inhibitory drugs; Rheumatoid arthritis; methotrexate
MeSH Terms: conditions — Hepatitis; Arthritis, Rheumatoid | interventions — Hepatitis A Vaccines; epaxal berna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: hepatitis A vaccine ( HAVRIX or EPAXAL) — 1.0 ml im ( Havrix) and 0.5 ml im (Epaxal. Both vaccines are given two times with 6 months interval

SUMMARY:
Hepatitis A vaccine is the most frequently used traveller's vaccine, yet data on its ability to induce protective immunity in immunosuppressed travellers are scarce. The investigators assess the hepatitis A virus (HAV) antibody response in patients with rheumatoid arthritis (RA) treated with Tumor Necrosis Factor (TNF) - inhibitors and/or methotrexate (Mtx).

DETAILED DESCRIPTION:
Methods: Parameters registered at baseline were: age, sex, duration of disease, medications, activity of disease (Visual Analogue Scale=VAS, Health Assessment Questionnaire Disability Index = HAQ, Disease Activity Score =DAS-28, CRP and total IgG in plasma). Hepatitis A vaccine (Epaxal or Havrix) were given at 0 and 6 months. Hepatitis A virus (HAV) antibodies is measured before vaccination and at month 1, 6 (before dose 2), 7 and 12 with quantitative HAV IgG, using the HAVAb-IgG Architect System, and by the HAVAB 2.0 assay on the AxSYM machine from Abbott. The level of protective immunity to HAV is defined as HAV IgG > 10mIU/mL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* TNF-alfa blocker and / or methotraxate in use as a medication against RA
* A desire to get protected against hepatitis A
* Men and women age 18-65 years
* Written informed consent
* Women of childbearing potential must use effective contraception -

Exclusion Criteria:

* Treatment with rituximab within 9 months before study start
* Known previous hepatitis A infection
* Previous vaccination against hepatitis A
* Allergy to eggs or formaldehyde
* Pregnancy or lactation
* Excessive use of alcohol
* Mental retardation
* Acute disease at the time of examination (fever > 38 degrees)
* Volunteer works as an employee of the researchers
* Previous vaccination against hepatitis A
* Egg-, henprotein- or formaldehyde allergy
* Pregnancy or lactation
* Excessive use of alcohol
* Another vaccine given within a month
* Acute disease at the time of examination (fever > 38 degrees)
* Not suitable for other reason in the investigator's opinion (other serious disease, i.e. AIDS/HIV-positive, cancer with ongoing cytostatic treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
seroconversion after a single dose of hepatitis A vaccine | one month after dose
  ELISA-titers are determined before first dose and at 1 and 6 months later

SECONDARY OUTCOMES:
seroconversion rates after a second dose of hepatitis A vaccine | 12 monrths
  We determine seroconversion rates before the second vaccine dose ( 6 months after the first) and at 1 and 6 months after the second dose

CONTACTS AND LOCATIONS:
Overall Officials: lars rombo, MD, Principal Investigator — Karolinska Institutet
Locations (4):
- Dept infectious diseases, Helsingfors, Finland
- Sweden (3):
  - Dept infectious diseases, Eskilstuna
  - Dept infectious diseases, Karlstad
  - Department of infectious diseases, Stockholm